CLINICAL TRIAL: NCT02136238
Title: A Clinical Trial Comparing Functional Performance of Voluntary Opening and Closing Body Powered Prosthetic Terminal Devices
Brief Title: Functional Performance of Voluntary Opening and Closing Body Powered Prostheses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: Florida High Tech Corridor Council (Other); TRS, Inc. (Industry)
Responsible Party: Principal Investigator, Jason Highsmith, Assistant Professor, University of South Florida
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Pro0013189
Record Dates: First submitted 2014-02-17; First posted 2014-05-12 (Estimated); Results first posted 2015-04-29 (Estimated); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Upper Limb Amputation
Keywords: amputation; transradial; prosthesis; terminal device

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Prosthetic hand 1 (Hosmer 5XA) (Active Comparator): This arm of the study included unilateral transradial amputees who who were assessed while using prosthetic hand 1
  Interventions: Device: Hosmer 5XA voluntary opening hook
- Prosthetic hand 2 (TRS Grip 3) (Active Comparator): This arm of the study included unilateral transradial amputees who who were assessed while using prosthetic hand 2
  Interventions: Device: TRS Grip 3 voluntary closing hook
- Non-amputee controls (No Intervention): This was an observational arm including non-amputees who were assessed as non-impaired control subjects. There are no interventions in this observational arm of the study.

INTERVENTIONS:
Device: Hosmer 5XA voluntary opening hook — Voluntary opening prosthetic terminal device ("hand")
  Arms: Prosthetic hand 1 (Hosmer 5XA)
Device: TRS Grip 3 voluntary closing hook — Voluntary closing prosthetic terminal device ("hand")
  Arms: Prosthetic hand 2 (TRS Grip 3)

SUMMARY:
This study will compare the functional performance of voluntary opening (VO) and voluntary closing (VC) body powered prostheses. We hypothesize that the ability to sense cable tension and produce progressively higher pinch from shoulder force will result in advantages for the VC terminal device (TRS, Grip 3) in terms of proprioception and overall function. The specific aims of this clinical trial are to:

1. Determine if accommodation with a VC Grip 3 prehensor will result in reduced compensatory motion during activity.
2. Determine if accommodation with a VC Grip 3 prehensor will result in improved function in activities of daily living.

DETAILED DESCRIPTION:
To evaluate the performance of the prehensors, subjects will complete a randomized A-B crossover study with a subjective follow-up. Two subject categories will be evaluated: 1.) healthy non-amputees, and 2.) unilateral transradial amputee subjects who currently use, or are interested in using a body-powered prosthesis. We anticipate data collection data with 10 non-amputee subject, and 8 amputee subjects.

ELIGIBILITY:
Inclusion criteria

* Unilateral transradial or wrist-disarticulation amputee
* 18 to 85 years of age
* At least 1 year from date of amputation
* Be able to independently provide informed consent
* Be willing to comply with study procedures Exclusion criteria
* History of acute or chronic skin breakdown on the residual limb
* Prosthetic socket adjustment within 90 days
* Any condition that would prevent participation and pose increased risk (e.g. shoulder impingement, sub-acromial bursitis, severe arthritis of the shoulder, elbow, wrist, or fingers)
* Injuries of the upper limb within the past 90 days (surgeries, sprains, strains, or fractures).
* Unwillingness/inability to follow instructions Inclusion criteria for able-bodied subjects
* 18 to 85 years of age
* Able to provide independent, informed consent
* Independent function by self-report
* Free of any health ailment that would impair physical function Exclusion criteria for able-bodied subjects
* Younger than 18 or older than 85 years of age
* Any condition that would prevent participation and pose increased risk (e.g. shoulder impingement, sub-acromial bursitis, severe arthritis of the shoulder, elbow, wrist, or fingers)
* No injuries of the upper limb within the past 90 days (surgeries, sprains, strains, or fractures).
* Unwillingness/inability to follow instructions

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-09; Primary Completion 2014-08 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Highsmith, PhD, Principal Investigator — University of South Florida
Locations (1):
- University of South Florida, Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Voluntary Open Device First Then Voluntary Close Device: Voluntary open device (Hosmer 5X hook terminal device) first then voluntary close device (TRS Grip 3 terminal device)
- Voluntary Close Device First Then Voluntary Open Device: Voluntary close device (TRS Grip 3 terminal device) first then voluntary open device (Hosmer 5X hook terminal device)
- Non-amputee Controls: This was an observational arm including non-amputees who were assessed as non-impaired control subjects. There are no interventions in this observational arm of the study.
  No intervention. Control group.: There are no interventions in this observational arm of the study.
Period: Overall Study
Arm/Group | Voluntary Open Device First Then Voluntary Close Device | Voluntary Close Device First Then Voluntary Open Device | Non-amputee Controls
Started | 4 | 4 | 10
Completed | 4 | 4 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Non-amputee Control Group: non-amputee healthy controls
- Experimental Group: Unilateral TR or Wrist-disartic Amputees: Includes groups randomized to receive either TRS Grip 3 voluntary close device or Hosmer 5XA voluntary open device first.
- Total: Total of all reporting groups
Arm/Group | Non-amputee Control Group | Experimental Group: Unilateral TR or Wrist-disartic Amputees | Total
Number analyzed (Participants) | 10 | 8 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.6 (6.0) | 56.1 (10.4) | 39.9 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 9 | 7 | 16
Region of Enrollment [Number; unit: participants]
  United States | 10 | 8 | 18

OUTCOME MEASURES:

1. Primary Outcome: Sternal Displacement During Towel Folding Task
Description: Distance sternum is displaced while folding a towel was measured in meters.
Time Frame: Based on preliminary experience with the intervention, accommodation can range from 1 month to 2 months. Assessment was scheduled within 1-2 weeks following accommodation.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Prosthetic Hand 1 (Hosmer 5XA) | Prosthetic Hand 2 (TRS Grip 3) | Non-amputee Controls
Number analyzed (Participants) | 8 | 8 | 10
meters | 1.0 (0.13) | 1.06 (0.12) | 0.88 (0.18)

2. Primary Outcome: Physical Function Performance 10 Test Score
Description: Simulation of 10 activities of daily living (i.e. donning a shirt, sweeping, walking stairs). Measured in units of time, distance and mass to provide a singular, continuous scaled score of function (from 0-100). A score of 100 is the maximal score and indicates the highest level of independent function where a score of 0 indicates the poorest score. Persons scoring lower scores will likely be at increased risk of dependency with daily function.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Voluntary Open (Hosmer 5XA): This arm of the study included unilateral transradial amputees who who were assessed while using prosthetic hand 1
- Voluntary Close (TRS Grip 3): This arm of the study included unilateral transradial amputees who who were assessed while using prosthetic hand 2
Arm/Group | Voluntary Open (Hosmer 5XA) | Voluntary Close (TRS Grip 3) | Non-amputee Controls
Number analyzed (Participants) | 8 | 8 | 10
units on a scale | 39.1 (13.5) | 37.0 (18.3) | 68.1 (14.2)

ADVERSE EVENTS:
Arm/Group | Voluntary Open (Hosmer 5XA) | Voluntary Close (TRS Grip 3) | Non-amputee Controls
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/10
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No